CLINICAL TRIAL: NCT07156760
Title: Morphological Characteristics of Spastic Musculature in the Upper and Lower Extremities Using Ultrasound Examination in Subjects After Stroke
Brief Title: Morphological Characteristics of the Upper and Lower Extremities Using Ultrasound Examination After Stroke.
Acronym: Spasticity
Status: Active, not recruiting | Type: Observational
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, ARLETTE PATRICIA DOUSSOULIN SANHUEZA, Associate professor, Universidad de La Frontera
Other Study IDs: DIUFRO FONDOS PROPIOS 240045; DIUFRO FONDOS PROPIOS 240045 (Registry Identifier: Morphological characteristics of spastic musculature)
Record Dates: First submitted 2025-08-10; First posted 2025-09-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: stroke; Spasticity Muscle; Ultrasound diagnostics
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound diagnostics — Non-invasive ultrasound evaluation of the upper limb on the hemiplegic side (Ekipomed Portable Ultrasound) to determine its pathological morphology (thickness, fiber orientation, and echogenicity) using the modified Heckmatt scale. This procedure will be performed by a physician who is an expert in muscle ultrasound.

SUMMARY:
Introduction A large number of stroke patients develop spasticity in the upper and lower extremities, which is one of the clinical signs of damage to motor neuron 1, causing abnormal postures and movement patterns due to motor neuron hyperexcitability and rheological alterations in the affected muscles. These alterations limit the use of the arm and leg, restricting their use in functional activities and affecting the quality of life and social participation of users. In recent years, the Heckmann scale has been used to evaluate spastic muscle alterations by ultrasound; however, evidence is limited regarding its benefits as an assessment tool for spastic hypertonia.

Objective To describe the morphological characteristics of spastic muscles in the lower extremities using ultrasound examination in subjects after stroke.

Method A prospective, multicenter descriptive study will be conducted. The sample will be non-probabilistic, consisting of 80 subjects who meet the eligibility criteria and provide informed consent.

Analysis of results Using the SPSS 27 program, a descriptive analysis will be performed using statistical indices of central tendency, dispersion, and distribution according to the measurement scale of each variable. The normality of the distribution of continuous variables will be investigated. In addition, a bivariate correlation analysis (ANOVA) will be performed. The significance level will be 0.05.

Expected Results It will provide updated evidence in the field of assessing the state of spastic muscles in subjects with neurological damage, a situation that will guide the therapeutic process and may improve the patient's prognosis and quality of life.

DETAILED DESCRIPTION:
Background: Spasticity is considered a positive clinical sign of upper motor neuron damage, associated with prevalent neurological pathologies such as stroke, constituting a clinical characteristic with a high incidence in the field of neurorehabilitation.

General Objective To describe the morphological characteristics of spastic biceps brachii and triceps surae muscles, using ultrasound examination, in subjects who have suffered a stroke.

Specific Objectives

1. Identify the morphological characteristics of the biceps, using ultrasound examination, in subjects after stroke.
2. Identify the morphological characteristics of the triceps surae, using ultrasound examination, in subjects after stroke.
3. Correlate the morphological characteristics of the biceps and triceps surae with the values obtained on the Ashworth and Tardieu scales.
4. Correlate the morphological characteristics of the biceps and triceps surae with the time of evolution and type of stroke.

Procedure

The first recruitment contact will be made by a professional from each participating center, who will inform the patient about the characteristics of the study and their future participation. Subsequently, eligibility criteria will be evaluated in order to identify 10 to 15 users per participating center.

After identification and signing of the consent form, participants will be invited to each center, where a professional will complete a structured clinical interview to obtain demographic and clinical data such as: type of stroke, time of onset, location, side affected, and treatments received.

Ultrasound evaluation Each participant will undergo a non-invasive ultrasound evaluation of the upper limb on the paralyzed side (using a portable Ekipomed ultrasound machine) to determine its pathological morphology (thickness, fiber orientation, and echogenicity) using the modified Heckmatt scale. This procedure will be performed by a physiatrist who is an expert in muscle ultrasound (with extensive experience and training in sonoanatomy). The technique involves placing the person in a supine or seated position, requesting that the biceps and triceps surae muscles be left free, then applying a colorless, hypoallergenic gel and proceeding with the examination by applying a transducer head to the gel located on the muscle to be evaluated. The procedure lasts 15 minutes per person.

nalysis All information will be compiled in an Excel database and statistically analyzed using SPSS 25 statistical software. The analysis will be descriptive, using statistical indices of central tendency, dispersion, and distribution according to the measurement scale of each variable. The normality of the distribution of continuous variables will be investigated. In addition, a bivariate correlation analysis will be performed using ANOVA. In all relevant analyses, the significance level will be 0.05.

Expected results Currently, advances in technology raise new questions and challenges. Given the above, this study will provide updated evidence in the field of neurorehabilitation assessment, associated with a pathology of high prevalence at the national and global level, such as stroke. This pathology manifests itself with clinical signs, including spastic hypertonia, a disorder that causes severe disability and affects people's quality of life. The results of this study will guide the therapeutic process, specifically in relation to the management of spastic hypertonia, a condition that can improve the patient's prognosis and promote a better quality of life and social interaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with a history of stroke more than three months ago.
* Who are undergoing or have undergone some type of rehabilitation in the acute and/or subacute stage.
* Who present spastic hypertonia in the upper and lower extremities detectable by Ashworth and Tardieu assessment.
* Presence of spastic pattern according to Hefter classification.
* Who agree to participate in the study and sign the consent form.

Exclusion Criteria:

* Structural joint involvement that prevents tone assessment.
* Patients who have been injected with antispastic drugs in the last 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult stroke patients with spasticity.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Spasticity | Outcome measure: Day 1, prior to the ultrasound scan. The results report will be issued 1 month after the analysis, sharing the analysis with participating centers and patients. On average, 1 year after the start of the study.
  Modified Ashworth Scale (MAS) The scale measures resistance during passive soft-tissue stretching. Lower values mean less spasticity
  Scoring:
  0 - No increase in muscle tone.
  1 - Slight increase in muscle tone, manifested by a catch and release at the end of the range of motion when the affected part(s) are moved in flexion or extension.
  1+ - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion.
  2 - More marked increase in muscle tone through most of the range of motion, but affected part(s) easily moved.
  3 - Considerable increase in muscle tone, passive movement difficult. 4 - Affected part(s) rigid in flexion or extension.

SECONDARY OUTCOMES:
Spasticity | Day 1, prior to the ultrasound scan. The results report will be issued 1 month after the analysis, sharing the analysis with participating centers and patients. On average, 1 year after the start of the study.
  Tardieu Scale (TS) Is a clinical tool used to assess spasticity by measuring the muscle's response to passive stretch at different velocities.
  The examiner moves the limb passively at three different speeds:
  V1: As slow as possible (to measure the full passive range of motion). V2: At the speed of the limb segment falling under gravity. V3: As fast as possible (faster than the natural drop of the limb under gravity).
  Two key measures are recorded:
  R1 (angle of catch): The angle at which a "catch" or resistance is first felt during a fast stretch.
  R2 (full passive range of motion): The angle of full joint range measured at slow speed.
  Interpretation:
  A large difference between R1 and R2 indicates a significant dynamic (neural) component of spasticity.
  A small difference suggests a greater fixed contracture or mechanical l
Morphological characteristics | Day 1, after the initial assessment. 5 patients per day, completing 15 per week at each center. Total intervention time, through study completion, an average of 6 months.
  The Modified Heckmatt Scale (MHS) is a clinical ultrasound grading system used to evaluate muscle echogenicity and architecture, particularly in patients with neuromuscular disorders. It assesses the degree of increased echogenicity (brightness) and loss of normal bone-muscle contrast, which reflect changes such as fibrosis, fatty infiltration, or atrophy.
  The scale typically ranges from Grade 1 (normal muscle: dark muscle with clear bone echo) to Grade 4 (severe abnormality: very bright muscle, bone echo poorly visible or lost).

CONTACTS AND LOCATIONS:
Overall Officials: Arlette P. Doussoulin, PhD, Principal Investigator — Universidad de La Frontera
Locations (2):
- Chile (2):
  - Universidad de La Frontera, Temuco, Región de la Araucanía
  - Universidad de La Frontera, Temuco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doussoulin A, Rivas R, Sabelle C. [Hospital discharges due to stroke in the period 2001-2010 in a southern Chilean region]. Rev Med Chil. 2016 May;144(5):571-6. doi: 10.4067/S0034-98872016000500003. Spanish. PMID 27552006
- [Background] Trompetto C, Marinelli L, Mori L, Pelosin E, Curra A, Molfetta L, Abbruzzese G. Pathophysiology of spasticity: implications for neurorehabilitation. Biomed Res Int. 2014;2014:354906. doi: 10.1155/2014/354906. Epub 2014 Oct 30. PMID 25530960
- [Background] Li S. Spasticity, Motor Recovery, and Neural Plasticity after Stroke. Front Neurol. 2017 Apr 3;8:120. doi: 10.3389/fneur.2017.00120. eCollection 2017. PMID 28421032